CLINICAL TRIAL: NCT04403451
Title: True North: Forging Pathways to Healthy Relationships and Economic Stability
Brief Title: True North Healthy Relationships Grant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Harbor, Inc. (Other)
Responsible Party: Principal Investigator, Dr. Leslie Leip, Principal Investigator, Children's Harbor, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90FM006902
Record Dates: First submitted 2017-07-18; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Behavior
Keywords: Relationships
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Experimental design with a randomized controlled trial for the impact evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1/Cohort 1 (Experimental): True North Love Notes, Financial Stability, Jobs
  Interventions: Behavioral: True North
- Phase 2/Cohort 2 (Experimental): True North Love Notes, Financial Stability, Jobs
  Interventions: Behavioral: True North
- Phase 3/Cohort 3 (Experimental): True North Love Notes, Financial Stability, Jobs
  Interventions: Behavioral: True North

INTERVENTIONS:
Behavioral: True North — Love Notes, Financial Stability, Jobs

SUMMARY:
The scientific purpose of the Children's Harbor True North evaluation study is to use a randomized controlled trial (RCT) to analyze the effects produced by True North and compare the outcomes of the program and comparison groups. The type of research for the RCT impact evaluation is behavioral.

The goal of the True North grant program is to successfully guide young adults who are randomly assigned to the program group through the transition from the foster care system to adulthood. The objectives of the True North program are to: 1) offer targeted, evidence-based healthy relationship interventions to the program group; 2) offer financial literacy to the program group in order for the participants to achieve greater economic stability; 3) provide job readiness sessions and connect the program group to subsidized and unsubsidized employment opportunities; and 4) match the young adults in the program group with a mentor to provide a permanent connection for guidance with relationship and financial issues.

The overall hypothesis is that participation in the True North program will increase the likelihood that the young adults will improve their relationships, improve their financial and employment stability, and improve their wellbeing.

DETAILED DESCRIPTION:
The investigator will use an experimental design using a randomized controlled trial for the impact evaluation of the True North program. This is a sound methodological design to assess the outcomes of the participants in the program and comparison groups. The target population is at-risk youth age 17 to 23 who have been involved in the foster care system and are preparing to "transition into adulthood." The units of analysis are young adults in the foster care system. The investigator plans to have 80-120 research study participants in each of the 3 cohorts. Over the 5-year grant period, a total of 300-360 young adults will be in the sample, with approximately 150-165 young adults in the program group and approximately 150-165 young adults in the comparison group. The inclusion criterion is: Any young adult age 17 to 23 who is aging out of the foster care system. The exclusion criterion does include an age restriction of 18 to 23 because that is the age group that receives extended foster care services in Broward County. Services end at age 24. There are no gender-based enrollment restrictions. There are no race-based enrollment restrictions.

The young adults randomly assigned to the program groups will take part in a multi-component intervention consisting of group workshops and individual sessions on relationship skills and financial stability and receive employment assistance and mentoring. For the healthy relationships component, program participants could receive 13 hours of workshops and 7 hours of individual sessions. For the economic stability component, program participants could receive 3.5 hours of financial stability and job readiness workshops and 7 hours of individual sessions about finance and employment. For the mentoring component, program participants could receive up to 7 hours of case management and 10 hours of prosocial events. All sessions will take place at the Children's Harbor Lauderhill office over a 9-month period.

The young adults in the program group will be completing a pre-test, post-test, and a followup. Answering the pre- and post-tests will take about 1 hour each and will be conducted at the Children's Harbor office, on the phone, or online. Participation in this evaluation study will take a total of approximately 106-112 hours of their time during the year-long program.

The investigator expects the True North program group to have improved relationship skills because of the participation in the Love Notes and mentoring components of the True North program. Love Notes v2.0, which was adapted from Relationships Smarts Plus, an evidence-based intervention rated by SAMSHA's National Registry of Evidence-based Programs and Practices (NREPP), will be utilized to help participants develop healthy relationship skills. It was selected based on its proven track record in serving diverse, economically disadvantaged youth and young adults age 16 to 24 who are at risk for poor quality relationships and unplanned pregnancies (NREPP 2012). An evaluation of Love Notes for Youth Build USA found that Love Notes participants improved their attitudes, knowledge, perceived skills, and behaviors associated with healthy relationships. When compared to with the control group, the Love Notes group had higher post program scores about their knowledge of healthy relationships.

The investigator expects True North participants to become financially stable through debt reduction, increased savings, improved credit scores, and asset building. The Annie E. Casey Foundation has developed a promising a practice of providing a coordinated set of services to help low-income individuals and families get jobs, strengthen their finances and move up the economic ladder. This practice entitled, Working Families Success Network (previously entitled the Center for Working Families), will be utilized to help participants develop financial literacy and job readiness skills. The Annie E. Casey Foundation reports that the Working Families Success Network model, which has been adopted at more than 100 locations throughout the country, has resulted in 4,400 people finding jobs, 3,300 getting steady 30-day employment, 2,300 obtaining public benefits, 2,800 improving their net worth, and 2,700 improving their credit score. Program participants also were five times more likely to achieve a major economic outcome - such as buying a car, getting out of debt or completing a training or education program - than the participants' counterparts who did not receive an intensive, coordinated set of services.

The True North program will support the development of job readiness skills, explore the participants' career interests, connect them to subsidized and unsubsidized job opportunities, and job coaching. The employment component will be supported by the True North Program Coordinator, Financial Coach, and Navigator. The Program Coordinator is developing relationships with employers to encourage and support job placement for participants. In addition, the Program Coordinator is working on implementing subsidized part time employment opportunities in the nonprofit arena. Participants will be prepared for these job opportunities by attending job readiness and career exploration sessions included in the financial literacy curriculum. The Financial Coach will also provide one-on-one job coaching as well as information on wages, benefits, and taxes. Most importantly, the participant's Navigator will guide the participants through a job hunt, provide support during the application and hiring process, and assist with job transitions.

ELIGIBILITY:
Inclusion Criteria:

* Young adult age 17 to 23
* Aging out of the foster care system in Broward County, Florida

Exclusion Criteria:

* Anyone not in foster care

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Healthy relationship measure from the Administration for Children and Families (ACF) Healthy Marriages post-program survey: "In a healthy relationship, it is essential for couples to talk about things that are important to them." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Higher score indicates better outcome.
Healthy relationship measure from the ACF Healthy Marriages post-program survey: "Even in a good relationship, couples will occasionally have trouble talking about their feelings." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Higher score indicates better outcome.
Healthy relationship measure from the ACF Healthy Marriages post-program survey: "A relationship is stronger if a couple doesn't talk about their problems." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Lower score indicates better outcome.
Job readiness measure from the ACF post-program survey: "You know where to find job openings." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Higher score indicates better outcome.
Job readiness measure from the ACF post-program survey: "You feel confident in your ability to conduct an effective job search for the job you want." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Higher score indicates better outcome.
Job readiness measure from the ACF post-program survey: "You know how to apply for a job." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Higher score indicates better outcome.
Job readiness measure from the ACF post-program survey: "You feel confident about your interviewing skills." | Immediately after the intervention
  4-point agreement scale (1=strongly disagree, 2=disagree, 3=agree, 4=strongly agree), Higher score indicates better outcome.
Financial assistance measure from the ACF follow-up survey: "Do you currently have enough income to cover regular expenses?" | Up to 24 weeks
  0=No, 1=Yes, Higher score indicates better outcome
Financial assistance measure from the ACF follow-up survey: "Do you currently have a checking account that you use?" | Up to 24 weeks
  0=No, 1=Yes, Higher score indicates better outcome
Financial assistance measure from the ACF follow-up survey: "Do you currently have a savings account?" | Up to 24 weeks
  0=No, 1=Yes, Higher score indicates better outcome
Financial assistance measure from the ACF follow-up survey: "Do you currently have money saved for an emergency?" | Up to 24 weeks
  0=No, 1=Yes, Higher score indicates better outcome
Life Satisfaction measure from National Accounts Measure of Well-being: "How satisfied are you with your life overall?" | Up to 24 weeks
  4-point satisfaction scale (1=very dissatisfied, 2=dissatisfied, 3=satisfied, 4=very satisfied), Higher score indicates a better outcome

SECONDARY OUTCOMES:
Relationship violence measure from the ACF Healthy Marriages post-program survey: "In a healthy relationship, how important is it that couples do not call each other names?" | Immediately after the intervention
  4-point importance scale (1=not at all important, 2=a little important, 3=pretty important, 4=very important), Higher score indicates better outcome.
Relationship violence measure from the ACF Healthy Marriages post-program survey: "In a healthy relationship, how important is it that couples do not threaten each other?" | Immediately after the intervention
  4-point importance scale (1=not at all important, 2=a little important, 3=pretty important, 4=very important), Higher score indicates better outcome.
Relationship violence measure from the ACF Healthy Marriages post-program survey: "In a healthy relationship, how important is it that couples do not push, shove, hit, slap or grab each other?" | Immediately after the intervention
  4-point importance scale (1=not at all important, 2=a little important, 3=pretty important, 4=very important), Higher score indicates better outcome.
Partner relationship measure from the ACF Healthy Marriages post-program survey: "How often do the following things happen with your partner/significant other - My partner can count on me to be there when he/she needs me." | Immediately after the intervention
  5-point scale (1=none of the time, 2=some of the time, 3=half of the time, 4=most of the time, 5= all of the time), Higher score indicates better outcome.
Partner relationship measure from the ACF Healthy Marriages post-program survey: "How often do the following things happen with your partner/significant other - My partner and I talk about things that really matter." | Immediately after the intervention
  5-point scale (1=none of the time, 2=some of the time, 3=half of the time, 4=most of the time, 5= all of the time), Higher score indicates better outcome.
Partner relationship measure from the ACF Healthy Marriages post-program survey: "How often do the following things happen with your partner/significant other - I am comfortable sharing my thoughts and feelings with my partner." | Immediately after the intervention
  5-point scale (1=none of the time, 2=some of the time, 3=half of the time, 4=most of the time, 5= all of the time), Higher score indicates better outcome.
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Do not have reliable transportation." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Do not have the right clothes." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Do not have documentation for legal employment." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Do not have good enough child care." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Have criminal record." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Do not have the education for good jobs." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Have substance abuse problem." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome
Employment measure from the ACF post-program survey: "How much does each of the following make it hard for you to find or keep a job? - Have mental health problem." | Immediately after the intervention
  3-point scale (1=never, 2=sometimes, 3=always), Lower score indicates better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Leip, Ph.D., Principal Investigator — Children's Harbor

IPD SHARING:
Plan to Share IPD: No